CLINICAL TRIAL: NCT01503112
Title: Does Urinary C-peptide Creatinine Ratio Predict Response to Incretin Based Agents in Type 2 Diabetes
Brief Title: Predicting Response to Incretin Based Agents in Type 2 Diabetes
Acronym: PRIBA
Status: Completed | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Exeter (Other)
Responsible Party: Principal Investigator, Angus Jones, NIHR Doctoral Research Fellow, Royal Devon and Exeter NHS Foundation Trust
Other Study IDs: 11233581
Record Dates: First submitted 2011-12-30; First posted 2012-01-02 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Type2 Diabetes
Keywords: Glucagon-Like Peptide 1, DPP4 protein, Therapeutics, Hypoglycemic Agents, C-Peptide, Type 2 Diabetes Mellitus,
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extracted DNA, stored serum/plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients starting incretin treatments: Patients starting GLP-1 agonists or DPPIV inhibitors as part of their normal clinical care.
  Interventions: Other: No intervention, observational study

INTERVENTIONS:
Other: No intervention, observational study

SUMMARY:
Type 2 diabetes is a major and rapidly increasing health problem worldwide. Keeping the blood glucose (sugar) from going too high helps prevent complications. Recently a number of new treatments (collectively called 'incretin based' treatments) to lower blood glucose have become available but response is very variable and it is difficult to predict which will work for an individual. The investigators want to see if we can identify whether the new treatments are likely to be effective for an individual patient. Identifying the right treatment would improve control and minimise the side-effects and costs from ineffective treatments. We will collect blood (for measures of blood glucose, insulin secretion and genetics information), urine (for a simple measurement of insulin secretion) and other clinical information (such as weight,age, duration of diabetes and medication) in people who are about to start these new 'incretin based' treatments and assess their response over the first 6 months of treatment. We will analyse this information to see if we can predict treatment response.

Study Hypothesis:

The investigators hypothesise that those who have low insulin secretion, as measured by post meal urine C-peptide Creatinine Ratio or blood C-peptide, will have poor blood glucose response to incretin based treatments.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of type 2 diabetes mellitus where the patient's clinician has determined the need for a DPP-IV inhibitor or GLP-1 analogue as a result of inadequate glycaemic control
* HbA1c >= 58mmol/mol

Exclusion Criteria:

* Treatment with DPP-IV inhibitors or GLP-1 analogues prior to study initiation (within the previous 3 months)
* Renal failure as shown by a eGFR (estimated glomerular filtration rate) less than 30 mL/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 Diabetes commencing DPP-IV inhibitors or GLP-1 agonsists in primary or secondary care in England
Sampling Method: Non-Probability Sample
Enrollment: 957 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Glycaemic response (HbA1c change post treatment) | 6 months
  Change in HbA1c over 6 months treatment (as a continuous variable and/or defined as binary response/non response). Our Primary analysis will be the relationship between insulin secretion (as measured by blood C-peptide or UCPCR) and glycaemic response. Secondary analysis will include examination of relationship between baseline weight, HbA1c, age, duration of diabetes, HOMA B, HOMA IR, autoantibody (GAD, IA2) status and glycaemic response. We will also examine the relationship between glycaemic response and polymorphisms in GLP-1R, TCF7L2, WFS1 and FOX01 genes.

SECONDARY OUTCOMES:
Weight change over 6 months treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Hattersley, Study Director — University of Exeter Medical School/Royal Devon and Exeter Hospital NHS Foundation Trust; Angus Jones, Principal Investigator — University of Exeter Medical School/Royal Devon and Exeter Hospital NHS Foundation Trust
Locations (18):
- United Kingdom (18):
  - Cornwall and Isles of Scilly NHS Primary Care Trust, Truro, Cornwall
  - North Devon NHS Trust, Barnstaple, Devon
  - Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon
  - Plymouth Hospitals NHS Trust, Plymouth, Devon
  - South Devon Healthcare NHS Foundation Trust, Torbay, Devon
  - Taunton and Somerset NHS Foundation Trust., Taunton, Somerset
  - Yeovil Disctrict Hospital NHS Foundation Trust, Yeovil, Somerset
  - The Royal Bournmouth and Christchurch Hospitals NHS Trust, Bournmouth
  - North Bristol NHS Trust, Bristol
  - Ipswich Hospital NHS Trust, Ipswich
  - Northampton General Hospital NHS Trust, Northampton
  - Oxford Radcliffe Hospitals NHS Trust, Oxford
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Surrey and Sussex Healthcare NHS trust, Redhill
  - East Sussex Healthcare NHS Trust, Saint Leonards-on-Sea
  - University Hospitls North Staffordshire NHS Trust, Stoke-on-Trent
  - South Warwickshire NHS Foundation Trust, Warwick
  - West Hertfordshire Hospitals NHS Trust, Watford

REFERENCES:
- [Result] Jones AG, McDonald TJ, Shields BM, Hill AV, Hyde CJ, Knight BA, Hattersley AT; PRIBA Study Group. Markers of beta-Cell Failure Predict Poor Glycemic Response to GLP-1 Receptor Agonist Therapy in Type 2 Diabetes. Diabetes Care. 2016 Feb;39(2):250-7. doi: 10.2337/dc15-0258. Epub 2015 Aug 4. PMID 26242184
- [Result] Dennis JM, Shields BM, Hill AV, Knight BA, McDonald TJ, Rodgers LR, Weedon MN, Henley WE, Sattar N, Holman RR, Pearson ER, Hattersley AT, Jones AG; MASTERMIND Consortium. Precision Medicine in Type 2 Diabetes: Clinical Markers of Insulin Resistance Are Associated With Altered Short- and Long-term Glycemic Response to DPP-4 Inhibitor Therapy. Diabetes Care. 2018 Apr;41(4):705-712. doi: 10.2337/dc17-1827. Epub 2018 Jan 31. PMID 29386249
- [Result] Jones AG, Shields BM, Hyde CJ, Henley WE, Hattersley AT. Identifying good responders to glucose lowering therapy in type 2 diabetes: implications for stratified medicine. PLoS One. 2014 Oct 23;9(10):e111235. doi: 10.1371/journal.pone.0111235. eCollection 2014. PMID 25340784
- See also: Research group website — http://www.diabetesgenes.org